CLINICAL TRIAL: NCT03054987
Title: Randomized Trial Comparing Endoscopic Ultrasound-guided Biliary Drainage (EUS-BD) and Endoscopic Retrograde Cholangiopancreatography (ERCP) for Malignant Distal Biliary Obstruction
Brief Title: Endoscopic Ultrasound and Endoscopic Retrograde Cholangiopancreatography for Malignant Distal Biliary Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 758636
Record Dates: First submitted 2017-01-17; First posted 2017-02-16 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Pancreatic Cancer; Pancreatic Neoplasms; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS-BD (Active Comparator): EUS-BD is a minimally invasive technique where the common bile duct (choledochoduodenostomy) is punctured under EUS-guidance and after transmural dilation, a stent is deployed for biliary drainage.
  Interventions: Procedure: EUS-BD
- ERCP (Active Comparator): At ERCP, the common bile duct will be selectively cannulated using a sphincterotome and guide wire technique. Once biliary access is obtained a stent will be deployed to facilitate biliary drainage.
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: EUS-BD — EUS-BD is a minimally invasive technique where the common bile duct (choledochoduodenostomy) is punctured under EUS-guidance and after transmural dilation, a stent is deployed for biliary drainage.
  Other Names: Endoscopic Ultrasound-guided biliary drainage
  Arms: EUS-BD
Procedure: ERCP — During the ERCP, a small catheter and guidewire is inserted into the bile duct and the stent can be deployed into the duct.
  Other Names: Endoscopic Retrograde Cholangiopancreatography
  Arms: ERCP

SUMMARY:
The purpose of this study is to compare the rates of adverse events between patients undergoing Endoscopic Ultrasound- guided biliary drainage and Endoscopic Retrograde Cholangiopancreatography for distal malignant biliary obstruction.

DETAILED DESCRIPTION:
The current curative treatment for patients with occlusion of the distal common bile duct by pancreatic cancer is pancreaticoduodenectomy (Whipple procedure). Unfortunately, more than 80% of patients have locally advanced or metastatic disease that requires neoadjuvant or palliative treatment. The goals of biliary drainage in the setting of locally advanced or metastatic pancreatic cancer are to palliate obstructive jaundice and lower serum bilirubin prior to systemic chemotherapy. In addition to resolving jaundice and associated pruritus, biliary drainage improves anorexia, indigestion and quality of life (1, 2). Endoscopic approach by means of retrograde cholangiopancreatography (ERCP) and biliary stent placement is the preferred treatment option for palliation of malignant obstructive jaundice. Endoscopic biliary drainage is safer than surgical bypass, with endoscopic placement of a plastic or metal stent having a lower relative risk of complications (3). When performed by experts, ERCP has favorable (80-90%) short-term (<90 days) success rates in the setting of malignant distal biliary obstruction (1-3). The rate of ERCP-associated adverse events (AEs) is 5-27% (4-7) and include pancreatitis, bleeding, infection, perforation and rarely death.

In a recent audit of 524 consecutive patients with an intact papilla who underwent ERCP at a tertiary endoscopy unit, 49 (9.4%) had a previously failed attempt at an outside facility and more than 80% of these failures were in the setting of a distal malignant stricture (8). Cancer in the pancreatic head or uncinate process can cause extensive ampullary inflammation that precludes successful biliary cannulation using standard techniques. In such circumstances, advanced techniques such as needle-knife sphincterotomy, dual wire technique, trans-papillary pancreatic sphincterotomy and cannulation over a pancreatic duct stent are performed to access the bile duct (9, 10). While the technical success rate for advanced techniques in expert hands is more than 85%, the procedure is associated with an AE rate of about 10-20% (9-11).

When ERCP is technically unsuccessful, patients are usually referred for interventional radiology-guided percutaneous transhepatic biliary drainage (PTBD). PTBD is usually a multi-step procedure that involves the initial placement of an external drainage catheter followed by internal trans-papillary stent placement. When the distal bile duct is severely strictured or when the intra-hepatic biliary system is non-dilated, PTBD is unsuccessful and is encountered in about 5-15% of patients with pancreatic cancer (12). The rate of short and long-term PTBD-related AEs is 5-10% and 20-30%, respectively (12-14). While most short-term AEs are due to infection and bleeding, the long-term AEs are due to stent dysfunction requiring frequent readmissions (12-14).

More recently, EUS-guided biliary drainage (EUS-BD) has emerged as a novel alternative to PTBD and ERCP for biliary decompression when advanced cannulation techniques fail. EUS-BD is a minimally invasive technique where the extra-hepatic common bile duct (choledochoduodenostomy) or intrahepatic bile duct (hepatogastrostomy) is punctured under EUS-guidance and after transmural dilation a stent is deployed for biliary drainage.

The potential advantages of EUS-BD are three-fold. Firstly, EUS-BD can be performed from multiple routes in the stomach and duodenum. Thus, duodenal stenosis is not a limitation to biliary access. Secondly, as biliary access is gained distant from the major duodenal papilla, the risk of post-procedure pancreatitis is low. Thirdly, as the deployed stent does not traverse the tumor, its patency could be longer. In a recent study of 95 patients with failed ERCP or inaccessible papilla, direct EUS-guided biliary drainage was successful in 86% of patients with an AE rate of 10.5% that included pancreatitis, bleeding, perforation, bile leak and infection (15). Most AEs were managed conservatively without the need for aggressive treatment measures. In another small, randomized trial of 25 patients with inoperable malignant biliary obstruction, there was no difference in clinical success, AEs, and costs between patients randomized to EUS-BD or PTBD (16). In a recent retrospective study of 208 patients with malignant obstructive jaundice treated by ERCP or EUS-BD directed biliary metal stent placement, there was no difference in the rates of technical success (>90% in both cohorts) or AEs (8.65% in both cohorts) between groups (17). However, patients who underwent ERCP had a 5% incidence of post-procedure pancreatitis compared to 0% in the EUS-BD cohort. Given these promising outcomes, EUS-BD is currently practiced as a complimentary therapy that allows biliary drainage when technical failure is encountered at ERCP. EUS-BD and PTBD have been shown to be comparable in effectiveness after failed ERCP, however patients who underwent PTBD had higher rates of adverse events and required additional interventions (19).

PTBD and EUS-BD have shown to be equally effective treatment options (16). The effectiveness of treatment outcomes between EUS-BD and ERCP needs to be evaluated. Since the treatment outcomes and safety profile of EUS-BD is comparable to ERCP and because EUS-BD is successful in more than 85% of patients with a failed ERCP, EUS-BD could be a first-line treatment option and not just a rescue measure for patients with malignant distal biliary obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Has jaundice due to malignant distal (more than 3cm distal to liver hilum) biliary obstruction.
3. The subject (or when applicable the subject's LAR) is able to understand and willing to sign an informed consent form prior to the initiation of any study procedures.

Exclusion Criteria:

1. Age <18 years
2. Females who are pregnant or lactating. Pregnancy in females of childbearing potential will be determined by routine preoperative urine HCG testing.
3. Coagulopathy which cannot be corrected (INR >1.6, thrombocytopenia with platelet count <50,000/ml)
4. Has surgically altered gastrointestinal anatomy such as but not limited to (Billroth II/Roux en-Y, gastric bypass).
5. Liver metastasis involving >30% of liver volume.
6. Liver cirrhosis with portal hypertension and/or ascites.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Rates of perforation | 1 week
  As defined by evidence of air or luminal contents outside the GI tract
Rates of pancreatitis | 1 week
  Defined as typical pain with amylase/lipase >3 times normal
Rates of bile leak | 1 week
  Not caused by pancreatitis or perforation
Rates of bleeding | 1 week
  As defined by "A lexicon for endoscopic adverse events: report of an ASGE workshop" PMID: 20189503
Rates of infection (cholangitis) | 1 week
  As defined by >38C >24 hours with cholestasis
Rates of peritionitis | 1 week
  As defined by "A lexicon for endoscopic adverse events: report of an ASGE workshop" PMID: 20189503
Rates of cholecystitis | 1 week
  As defined by "A lexicon for endoscopic adverse events: report of an ASGE workshop" PMID: 20189503
Rates of pneumoperitoneum | 1 week
  As defined by "A lexicon for endoscopic adverse events: report of an ASGE workshop" PMID: 20189503
Rates of fever | 1 week
  Defined as temperature >38C
Rates of abdominal pain | 1 week
  Defined as pain described by the patient not caused by pancreatitis or perforation
Rates of death attributable to the procedure. | 1 week
  As defined by "A lexicon for endoscopic adverse events: report of an ASGE workshop" PMID: 20189503

SECONDARY OUTCOMES:
Technical Success | 1 day
  Defined as successful placement of a stent for malignant distal biliary obstruction in the desired location as determined at ERCP and EUS in the index session.
Treatment success | 2 weeks
  Clinical success is defined as decrease in direct bilirubin by 50% at 2 weeks
Procedural duration | 1 day
  Defined as the time between procedure onset and completion of the procedure (stent deployment). The duration will be calculated in minutes from the time the echoendoscope or duodenoscope is positioned and the stent is deployed.
Reintervention | 6 months
  Need for additional intervention (endoscopic, surgical or radiological) to relieve jaundice in the presence of dilated biliary system

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Center for Interventional Endoscopy - Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared via publication and/or presentation.
Supporting Information: SAP

REFERENCES:
- [Background] Barkay O, Mosler P, Schmitt CM, Lehman GA, Frakes JT, Johanson JF, Qaseem T, Howell DA, Sherman S. Effect of endoscopic stenting of malignant bile duct obstruction on quality of life. J Clin Gastroenterol. 2013 Jul;47(6):526-31. doi: 10.1097/MCG.0b013e318272440e. PMID 23269313
- [Background] Pereira-Lima JC, Jakobs R, Maier M, Kohler B, Benz C, Martin WR, Riemann JF. Endoscopic stenting in obstructive jaundice due to liver metastases: does it have a benefit for the patient? Hepatogastroenterology. 1996 Jul-Aug;43(10):944-8. PMID 8884318
- [Background] Moss AC, Morris E, Mac Mathuna P. Palliative biliary stents for obstructing pancreatic carcinoma. Cochrane Database Syst Rev. 2006 Apr 19;2006(2):CD004200. doi: 10.1002/14651858.CD004200.pub4. PMID 16625598
- [Background] Coelho-Prabhu N, Shah ND, Van Houten H, Kamath PS, Baron TH. Endoscopic retrograde cholangiopancreatography: utilisation and outcomes in a 10-year population-based cohort. BMJ Open. 2013 May 31;3(5):e002689. doi: 10.1136/bmjopen-2013-002689. PMID 23793659
- [Background] Lee JH, Krishna SG, Singh A, Ladha HS, Slack RS, Ramireddy S, Raju GS, Davila M, Ross WA. Comparison of the utility of covered metal stents versus uncovered metal stents in the management of malignant biliary strictures in 749 patients. Gastrointest Endosc. 2013 Aug;78(2):312-24. doi: 10.1016/j.gie.2013.02.032. Epub 2013 Apr 13. PMID 23591331
- [Background] Andriulli A, Loperfido S, Napolitano G, Niro G, Valvano MR, Spirito F, Pilotto A, Forlano R. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol. 2007 Aug;102(8):1781-8. doi: 10.1111/j.1572-0241.2007.01279.x. Epub 2007 May 17. PMID 17509029
- [Background] Williams EJ, Taylor S, Fairclough P, Hamlyn A, Logan RF, Martin D, Riley SA, Veitch P, Wilkinson ML, Williamson PR, Lombard M. Risk factors for complication following ERCP; results of a large-scale, prospective multicenter study. Endoscopy. 2007 Sep;39(9):793-801. doi: 10.1055/s-2007-966723. PMID 17703388
- [Background] Holt BA, Hawes R, Hasan M, Canipe A, Tharian B, Navaneethan U, Varadarajulu S. Biliary drainage: role of EUS guidance. Gastrointest Endosc. 2016 Jan;83(1):160-5. doi: 10.1016/j.gie.2015.06.019. Epub 2015 Jul 26. PMID 26215648
- [Background] Swan MP, Alexander S, Moss A, Williams SJ, Ruppin D, Hope R, Bourke MJ. Needle knife sphincterotomy does not increase the risk of pancreatitis in patients with difficult biliary cannulation. Clin Gastroenterol Hepatol. 2013 Apr;11(4):430-436.e1. doi: 10.1016/j.cgh.2012.12.017. Epub 2013 Jan 11. PMID 23313840
- [Background] Glomsaker T, Hoff G, Kvaloy JT, Soreide K, Aabakken L, Soreide JA; Norwegian Gastronet ERCP Group. Patterns and predictive factors of complications after endoscopic retrograde cholangiopancreatography. Br J Surg. 2013 Feb;100(3):373-80. doi: 10.1002/bjs.8992. Epub 2012 Dec 6. PMID 23225493
- [Background] Kahaleh M, Tokar J, Mullick T, Bickston SJ, Yeaton P. Prospective evaluation of pancreatic sphincterotomy as a precut technique for biliary cannulation. Clin Gastroenterol Hepatol. 2004 Nov;2(11):971-7. doi: 10.1016/s1542-3565(04)00484-7. PMID 15551249
- [Background] Crosara Teixeira M, Mak MP, Marques DF, Capareli F, Carnevale FC, Moreira AM, Ribeiro U Jr, Cecconello I, Hoff PM. Percutaneous transhepatic biliary drainage in patients with advanced solid malignancies: prognostic factors and clinical outcomes. J Gastrointest Cancer. 2013 Dec;44(4):398-403. doi: 10.1007/s12029-013-9509-3. PMID 23760941
- [Background] Zhang GY, Li WT, Peng WJ, Li GD, He XH, Xu LC. Clinical outcomes and prediction of survival following percutaneous biliary drainage for malignant obstructive jaundice. Oncol Lett. 2014 Apr;7(4):1185-1190. doi: 10.3892/ol.2014.1860. Epub 2014 Feb 7. PMID 24944690
- [Background] Lee E, Gwon DI, Ko GY, Sung KB, Yoon HK, Shin JH, Kim JH, Ko HK, Song HY. Percutaneous biliary covered stent insertion in patients with malignant duodenobiliary obstruction. Acta Radiol. 2015 Feb;56(2):166-73. doi: 10.1177/0284185114523267. Epub 2014 Feb 11. PMID 24518689
- [Background] Shah JN, Marson F, Weilert F, Bhat YM, Nguyen-Tang T, Shaw RE, Binmoeller KF. Single-operator, single-session EUS-guided anterograde cholangiopancreatography in failed ERCP or inaccessible papilla. Gastrointest Endosc. 2012 Jan;75(1):56-64. doi: 10.1016/j.gie.2011.08.032. Epub 2011 Oct 21. PMID 22018554
- [Background] Artifon EL, Aparicio D, Paione JB, Lo SK, Bordini A, Rabello C, Otoch JP, Gupta K. Biliary drainage in patients with unresectable, malignant obstruction where ERCP fails: endoscopic ultrasonography-guided choledochoduodenostomy versus percutaneous drainage. J Clin Gastroenterol. 2012 Oct;46(9):768-74. doi: 10.1097/MCG.0b013e31825f264c. PMID 22810111
- [Background] Dhir V, Itoi T, Khashab MA, Park DH, Yuen Bun Teoh A, Attam R, Messallam A, Varadarajulu S, Maydeo A. Multicenter comparative evaluation of endoscopic placement of expandable metal stents for malignant distal common bile duct obstruction by ERCP or EUS-guided approach. Gastrointest Endosc. 2015 Apr;81(4):913-23. doi: 10.1016/j.gie.2014.09.054. Epub 2014 Dec 5. PMID 25484326
- [Background] Khashab MA, Valeshabad AK, Afghani E, Singh VK, Kumbhari V, Messallam A, Saxena P, El Zein M, Lennon AM, Canto MI, Kalloo AN. A comparative evaluation of EUS-guided biliary drainage and percutaneous drainage in patients with distal malignant biliary obstruction and failed ERCP. Dig Dis Sci. 2015 Feb;60(2):557-65. doi: 10.1007/s10620-014-3300-6. Epub 2014 Aug 1. PMID 25081224
- [Result] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Derived] Bang JY, Navaneethan U, Hasan M, Hawes R, Varadarajulu S. Stent placement by EUS or ERCP for primary biliary decompression in pancreatic cancer: a randomized trial (with videos). Gastrointest Endosc. 2018 Jul;88(1):9-17. doi: 10.1016/j.gie.2018.03.012. Epub 2018 Mar 21. PMID 29574126